CLINICAL TRIAL: NCT06535958
Title: Impact of Oral Hygiene Instructions in the Resolution of Peri-implant Mucositis. A Randomized Clinical Trial
Brief Title: Impact of Oral Hygiene Instructions in the Resolution of Peri-implant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Beatriz de Tapia, Assistant professor, Department of Periodontology, Universitat Internacional de Catalunya (UIC), Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER-ECL-2023-07
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (OHI) (Experimental)
  Interventions: Behavioral: OHI
- Control Group (OHI+PMPR) (Experimental)
  Interventions: Behavioral: OHI; Procedure: OHI+PMPR

INTERVENTIONS:
Behavioral: OHI — All patients (test and control) will be instructed to brush the implants twice daily to remove supragingival biofilms with a low-abrasive dentifrice and to use specific cylindrical or conical brushes in the interproximal area. Patients will be indicated to brush under, around, and in the peri-implant crevice circumferentially. In those cases with no access for proper OHI, prosthesis will be modified.The interproximal brush device used will be chosen for the patient individually, according to the interproximal space available, the thicker brush that can be used comfortably will be the selected one. It will be previously tested on the patient and its use will be taught, patients should demonstrate proficiency
Procedure: OHI+PMPR — Supra- and sub-gingival debridement of the implant surface, the implant neck, and the abutment will be carried out by means of a combination of ultrasonics with a plastic tip and plastic curettes . Finally, the prosthetic components will be polished with a rubber cup
  Arms: Control Group (OHI+PMPR)

SUMMARY:
Peri-implant mucositis (PM) over dental implants is a highly prevalent disease characterized by inflammation of the peri-implant mucosa without loss of supporting bone around implants. If untreated, PM may progress into peri-implantitis, which may ultimately lead to implant loss. Multiple clinical studies have described a cause-effect relationship between the accumulation of biofilm and the development of PM and therefore effective oral hygiene practices and professional biofilm control are fundamental in their prevention and management. As it was stated in the latest expert consensus on the prevention and treatment of peri-implant diseases, up to date, the treatment of PM includes mechanical professional cleaning associated with oral hygiene instructions (OHI). However, the impact of OHI by itself is not known. This randomized clinical trial over 56 patients aims to identify if there is any superiority of individualized OHI and mechanical/physical instrumentation over OHI alone. The main objective is to evaluate the resolution of the disease, by means of reduction of modified bleeding index (mBI) 1 and 3 months after treatment. Secondary objectives include evaluating microbiological changes and determining if the extent of inflammation measured as the initial mBI could have any impact on PM resolution after different treatment modalities.In addition, the hypotheses formulated are as follows;

* The proper oral hygiene measures conducted by the patient after individualized OHI will achieve resolution of PM in a clinically relevant proportion of patients.
* The proper oral hygiene measures conducted by the patient after individualized OHI will reduce the expression of peri-implant pathogens as much as the combination of individualized OHI and professional mechanical debridement in a clinically relevant proportion of patients.
* The proper oral hygiene measures conducted by the patient after individualized OHI will reduce mBI as much as the combination of individualized OHI and professional mechanical debridement in a clinically relevant proportion of patients.
* The extent of inflammation measured as the mBI could be related with the degree of resolution of the disease according to the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of, at least, one titanium implant that have been more than one year in function and exhibits PM, defined as bleeding on gentle probing (0.20 N) in at least one peri-implant site.
2. No signs of loss of supporting bone after initial bone remodelling. In cases where baseline radiograph is available, it will be used for comparison, otherwise a maximum of 2 mm of crestal bone loss will be accepted
3. Presence of >1 mm of keratinized peri-implant mucosa.
4. Absence of systemic diseases that could influence the outcome of the therapy (i.e. controlled diabetes, with HbA1c<7, patients will be included).
5. Non-smoker or light smoking status in smokers (<10 cigarettes/day)

Exclusion Criteria:

1. Untreated periodontal conditions.
2. Pregnant or lactating women.
3. Patients who received systemic antibiotics in the last 3 months.
4. Patients who received treatment of PM in the past 3 months.
5. Patients receiving corticoids or medications known to have effect on gingival growth (i.e., calcium channel antagonists, immunosuppressants or antiepileptic drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Modified bleeding index | At baseline, 1 and 3 months after treatment
  An electronic pressure-calibrated probe is used. The index is measured tooth by tooth, and later averaged. The minimum value is 0 and the maximum value is 3, with the best value being 0 and the worst value being 3.

SECONDARY OUTCOMES:
Full mouth plaque Index | At baseline, 1 and 3 months after treatment
  A periodontal probe is used. Assessed dichotomously at four sites per tooth (mesial, buccal, distal, and lingual); 1 meaning presence of plaque and 0 abscense. This index is measured by the percentage of sites with plaque over the total number of sites evaluated.
Full mouth bleeding index | At baseline, 1 and 3 months after treatment
  Electronic pressure-calibrated probe. Assessed dichotomously as presence or absence of bleeding after 30 seconds of gently probing.1 meaning presence of blood and 0 abscense This index is measured by the percentage of sites bleeding over the total number of sites evaluated.
Full mouth probing pocket depth | At baseline, 1 and 3 months after treatment
  Electronic pressure-calibrated probe. Measured at six sites around each tooth, except third molars. Is used to measure the millimeters that the probe is introduced through the gingival sulcus.
Suppuration on probing | At baseline, 1 and 3 months after treatment
  Electronic pressure-calibrated probe. Assessed dichotomously as presence or absence of suppuration within 30 seconds after probing. 1 meaning presence of suppuration and 0 abcense
Implant probing pocket depth | At baseline, 1 and 3 months after treatment
  Electronic pressure-calibrated probe. This index is used to know the millimeters that the probe is introduced through the peri-implant sulcus.
Microbiological test | At baseline, 1 and 3 months after treatment.
  Sterile paper points. Detect the absence or presence of certain types of bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz de Tapia Pastor, DDS,MSC,PhD, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Sant Cugat Del Vallès, Spain

IPD SHARING:
Plan to Share IPD: Yes
The results obtained are expected to be published in both national and international journals. In addition, the results will be disseminated national and international scientific events.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT06535958/Prot_SAP_000.pdf